CLINICAL TRIAL: NCT00448110
Title: Randomized, Double-Blind, Active- and Placebo-Controlled Study of the Efficacy and Safety of Repeated Dosing of DIC075V Relative To Parenteral Ketorolac and Placebo in Patients With Acute Post-Op Pain After Abdominal or Pelvic Surgery
Brief Title: Efficacy and Safety of IV Diclofenac (DIC075V) for Pain After Abdominal or Pelvic Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Javelin Pharmaceuticals (Industry)
Responsible Party: Javelin Pharmaceuticals, Javelin Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DFC-004
Record Dates: First submitted 2007-03-13; First posted 2007-03-15 (Estimated); Last update posted 2009-05-22 (Estimated); Status verified 2009-05

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- A (Experimental): intravenous diclofenac dosage level 1
  Interventions: Drug: Intravenous Diclofenac (DIC075V)
- B (Experimental): intravenous diclofenac dosage level 2
  Interventions: Drug: Intravenous Diclofenac (DIC075V)
- C (Active Comparator): intravenous ketorolac
  Interventions: Drug: Intravenous Ketorolac
- D (Placebo Comparator): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Intravenous Diclofenac (DIC075V) — Intravenous Diclofenac (DIC075V): 1 of 2 dosage levels
  Arms: A; B
Drug: Intravenous Ketorolac — Intravenous Ketorolac
  Arms: C
Drug: placebo — placebo
  Arms: D

SUMMARY:
This study will compare repeated intermittent IV dosing of diclofenac in patients with moderate to severe post-surgical pain from abdominal or pelvic surgery.

DETAILED DESCRIPTION:
The primary objective is to evaluate the efficacy and safety of two dosage levels of parenteral diclofenac in providing pain relief as compared to placebo or Ketorolac tromethamine.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled within two weeks of the screening visit to undergo abdominal or pelvic surgery
* Moderate to severe pain within 6 hours following completion of the required surgery.

Exclusion Criteria:

* Surgical procedure involves a subcostal incision.
* Chronic disease or recent cardiovascular events.
* Known allergy or hypersensitivity to the active compounds or any of the excipients used in the study.

Additional Inclusion/Exclusion Criteria May Apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 331 (Actual)
Dates: Start 2006-05; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Sum of the pain intensity differences (SPID) over the 0-48 hour time interval. | 0-48 hours

SECONDARY OUTCOMES:
SPID over the 0-24 hour interval | 0-24 hours
Other measures of pain relief | Multiple

CONTACTS AND LOCATIONS:
Overall Officials: Javelin Pharmaceuticals, Study Director — Javelin Pharmaceuticals
Locations (14):
- United States (14):
  - Alabama Clinical Therapeutics, Birmingham, Alabama
  - Eliza Coffee Memorial Hospital, Florence, Alabama
  - Drug Research and Analysis Corp., Montgomery, Alabama
  - Helen Keller Hospital, Sheffield, Alabama
  - Teton Research / Parkview Surgical, Little Rock, Arkansas
  - Glendale Adventist Medical Center, Glendale, California
  - Saddleback Memorial Medical Center, Laguna Hills, California
  - Visions Clinical Research, Boynton Beach, Florida
  - Duke University Medical Center, Durham, North Carolina
  - Clinical Research Services, Bismarck, North Dakota
  - Clinical Research Center, Austin, Texas
  - Memorial Hermann Healthcare System - Memorial City Hospital, Houston, Texas
  - Clinical Research Center, San Marcos, Texas
  - Jean Brown Research, Salt Lake City, Utah

REFERENCES:
- [Derived] Chelly JE, Lacouture PG, Reyes CRD. Safety of Injectable HPbetaCD-Diclofenac in Older Patients with Acute Moderate-to-Severe Postoperative Pain: A Pooled Analysis of Three Phase III Trials. Drugs Aging. 2018 Mar;35(3):249-259. doi: 10.1007/s40266-018-0529-3. PMID 29492863
- [Derived] Gan TJ, Daniels SE, Singla N, Hamilton DA, Carr DB. A novel injectable formulation of diclofenac compared with intravenous ketorolac or placebo for acute moderate-to-severe pain after abdominal or pelvic surgery: a multicenter, double-blind, randomized, multiple-dose study. Anesth Analg. 2012 Nov;115(5):1212-20. doi: 10.1213/ANE.0b013e3182691bf9. Epub 2012 Aug 10. PMID 22886837